CLINICAL TRIAL: NCT02597036
Title: A Phase 1 Study of LY3127804 as Monotherapy and in Combination With Ramucirumab in Patients With Advanced Solid Tumors
Brief Title: A Study of LY3127804 With Ramucirumab in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15580; I7W-MC-JQBA (Other: Eli Lilly and Company); 2015-001204-64 (EudraCT Number)
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors
Keywords: Advanced, Angiopoietin
MeSH Terms: interventions — zansecimab; Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part A LY3127804 (Experimental): Participants received escalating doses of 4 milligram per kilogram (mg/kg), 8 mg/kg, 12 mg/kg, 16 mg/kg, 20 mg/kg and 27 mg/kg LY3127804 administered as intravenous (IV) infusion on days 1 and 15 of a 28-day cycle.
  Interventions: Drug: LY3127804
- Part B LY3127804 + 8 mg/kg Ramucirumab (Experimental): Participants received escalating doses of 8 mg/kg / 12 mg/kg / 16 mg/kg / 20 mg/kg / 27 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
  Interventions: Drug: LY3127804; Drug: Ramucirumab
- Part C LY3127804 + 12 mg/kg Ramucirumab (Experimental): Participants received 20 mg/kg LY3127804 plus 12 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
  Interventions: Drug: LY3127804; Drug: Ramucirumab
- Part D LY3127804 + Ramucirumab - Not Enrolled (Experimental): Participants were to receive LY3127804 and Ramucirumab IV Q2W until participant qualifies for study discontinuation.
  Part D and E were not enrolled based on the primary and secondary outcomes/ results of Part A-C.
  Interventions: Drug: LY3127804; Drug: Ramucirumab
- Part E LY3127804 + Ramucirumab + Paclitaxel - Not Enrolled (Experimental): Participants were to receive LY3127804 and Ramucirumab IV Q2W and Paclitaxel IV on day 1, 8, and 15 until participant qualifies for study discontinuation.
  Part D and E were not enrolled based on the primary and secondary outcomes/ results of Part A-C.
  Interventions: Drug: LY3127804; Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: LY3127804 — Administered IV
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806; Cyramza; 1121B
  Arms: Part B LY3127804 + 8 mg/kg Ramucirumab; Part C LY3127804 + 12 mg/kg Ramucirumab; Part D LY3127804 + Ramucirumab - Not Enrolled; Part E LY3127804 + Ramucirumab + Paclitaxel - Not Enrolled
Drug: Paclitaxel — Administered IV
  Arms: Part E LY3127804 + Ramucirumab + Paclitaxel - Not Enrolled

SUMMARY:
The main purpose of this study is to evaluate the safety of the study drug known as LY3127804 given as monotherapy and in combination with Ramucirumab for participants with advanced or metastatic solid tumors. The study will also include a safety exploration for the combination of LY3127804 plus ramucirumab and paclitaxel

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cancer that is advanced and/or metastatic.
* Have disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST ) version 1.1.
* Have adequate organ function.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Have discontinued previous treatments for cancer for at least 28 days or 5 half-lives prior to study enrolment.

Exclusion Criteria:

* Have serious preexisting medical conditions.
* Have received treatment with a drug predominantly targeting Ang2 activity.
* Have symptomatic central nervous system (CNS) malignancy or metastasis.
* Have current hematologic malignancies.
* Have an active fungal, bacterial, and/or known viral infection.
* Have a corrected QT interval using Fridericia's correction (QTcF) of >470 msec on screening electrocardiogram (ECG) at several consecutive days of assessment.
* Have a known sensitivity to mAbs or other therapeutic proteins.
* Have a history of hypertensive crisis or hypertensive encephalopathy or current poorly controlled hypertension despite standard medical management.
* Have a significant bleeding disorder or vasculitis or had a Grade ≥3 bleeding episode within 3 months prior to receiving treatment.
* Receive anticoagulation therapy at therapeutic dose.
* Have experienced any arterial or venothrombotic or thromboembolic events within 6 months prior to study treatment.
* Have liver cirrhosis with a Child-Pugh class B or worse or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis.
* The participant is pregnant prior to randomization or breastfeeding.
* The participant has sensory peripheral neuropathy ≥ Grade 2 (Part E only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2020-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (2):
  - SMO Sarah Cannon Research Inst., Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels, Belgium
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villejuif, France
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona, Spain

REFERENCES:
- [Derived] Martin-Liberal J, Hollebecque A, Aftimos P, Jungels C, Martin-Romano P, Rodon J, Kremer JD, Zhang W, Bendell J. First-in-human, dose-escalation, phase 1 study of anti-angiopoietin-2 LY3127804 as monotherapy and in combination with ramucirumab in patients with advanced solid tumours. Br J Cancer. 2020 Oct;123(8):1235-1243. doi: 10.1038/s41416-020-1011-7. Epub 2020 Aug 3. PMID 32741971
- See also: A Study of LY3127804 with Ramucirumab in Participants with Advanced Solid Tumors — https://trials.lillytrialguide.com/en-US/trial/3wy8LzQ4ukMaWSwg8k8OaW

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are participants that completes cycle 1 (28 Day Cycle).
Groups:
- Part A Cohort 1: 4 Milligram Per Kilogram (mg/kg) LY3127804: Participants received 4 mg/kg LY3127804 administered as intravenous (IV) infusion on days 1 and 15 of a 28-day cycle.
- Part A Cohort 2: 8 mg/kg LY3127804: Participants received 8 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part A Cohort 3: 12 mg/kg LY3127804: Participants received 12 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part A Cohort 4: 16 mg/kg LY3127804: Participants received 16 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part A Cohort 5: 20 mg/kg LY3127804: Participants received 20 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part A Cohort 6: 27 mg/kg LY3127804: Participants received 27 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part B Cohort 2: 8 mg/kg LY3127804 + 8 mg/kg Ramucirumab: Participants received 8 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part B Cohort 3: 12 mg/kg LY3127804 + 8 mg/kg Ramucirumab: Participants received 12 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part B Cohort 4: 16 mg/kg LY3127804 + 8 mg/kg Ramucirumab: Participants received 16 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part B Cohort 5: 20 mg/kg LY3127804 + 8 mg/kg Ramucirumab: Participants received 20 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part B Cohort 6: 27 mg/kg LY3127804 + 8 mg/kg: Participants received 27 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part C: 20 mg/kg LY3127804 +12 mg/kg Ramucirumab: Participants received 20 mg/kg LY3127804 plus 12 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
Period: Overall Study
Arm/Group | Part A Cohort 1: 4 Milligram Per Kilogram (mg/kg) LY3127804 | Part A Cohort 2: 8 mg/kg LY3127804 | Part A Cohort 3: 12 mg/kg LY3127804 | Part A Cohort 4: 16 mg/kg LY3127804 | Part A Cohort 5: 20 mg/kg LY3127804 | Part A Cohort 6: 27 mg/kg LY3127804 | Part B Cohort 2: 8 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 3: 12 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 4: 16 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 5: 20 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 6: 27 mg/kg LY3127804 + 8 mg/kg | Part C: 20 mg/kg LY3127804 +12 mg/kg Ramucirumab
Started | 3 | 4 | 3 | 3 | 3 | 4 | 6 | 7 | 7 | 7 | 8 | 7
Received at Least 1 Dose of Study Drug | 3 | 4 | 3 | 3 | 3 | 4 | 6 | 7 | 7 | 7 | 8 | 7
Completed | 3 | 4 | 3 | 3 | 2 | 3 | 5 | 6 | 7 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 2
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants in Part A, Part B and Part C.
Groups:
- Part A Cohort 1: 4 mg/kg LY3127804: Participants received 4 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1: 4 mg/kg LY3127804 | Part A Cohort 2: 8 mg/kg LY3127804 | Part A Cohort 3: 12 mg/kg LY3127804 | Part A Cohort 4: 16 mg/kg LY3127804 | Part A Cohort 5: 20 mg/kg LY3127804 | Part A Cohort 6: 27 mg/kg LY3127804 | Part B Cohort 2: 8 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 3: 12 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 4: 16 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 5: 20 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 6: 27 mg/kg LY3127804 + 8 mg/kg | Part C: 20 mg/kg LY3127804 +12 mg/kg Ramucirumab | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 4 | 6 | 7 | 7 | 7 | 8 | 7 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.30 (11.72) | 54.30 (7.80) | 58.70 (13.05) | 66.00 (5.57) | 66.00 (15.13) | 62.80 (10.72) | 57.80 (9.41) | 55.30 (12.65) | 51.90 (19.58) | 65.60 (6.53) | 50.60 (12.11) | 54.40 (9.13) | 57.30 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 1 | 3 | 3 | 3 | 1 | 2 | 1 | 5 | 3 | 26
  Male | 2 | 2 | 2 | 2 | 0 | 1 | 3 | 6 | 5 | 6 | 3 | 4 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 3 | 2 | 2 | 4 | 3 | 6 | 6 | 5 | 6 | 5 | 45
  Unknown or Not Reported | 2 | 2 | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 2 | 1 | 2 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 4
  White | 1 | 4 | 3 | 3 | 3 | 3 | 6 | 7 | 4 | 7 | 8 | 7 | 56
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 3 | 1 | 1 | 3 | 1 | 15
  France | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 3 | 2 | 0 | 3 | 17
  Spain | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 1 | 12
  United States | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 2 | 2 | 3 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose of LY3127804 Monotherapy and in Combination With Ramucirumab
Description: Recommended Phase 2 dose was determined based on observed safety, pharmacokinetics (PK) and efficacy. However maximum tolerated dose (MTD) was not determined. For the purpose of this study, the MTD is defined as the highest tested dose in a single-agent setting that has less than (<) 33% probability of causing a DLT. MTD in the combination setting was determined based on the nature and timing of the DLTs in the combination setting. Dose-limiting toxicities were not reported in any treatment cohort. Therefore, the maximum tolerated LY3127804 dose could not be determined.
Time Frame: Baseline through Cycle 1 (28 Day Cycle)
Population: All randomized participants who received at least one dose of study drug (ramucirumab and/or LY3127804) in Part A, Part B and Part C.
Measure: Number; unit: milligram per kilogram (mg/kg)
Groups:
- All Part A , Part B and Part C Participants: Part A: Participants received escalating doses of 4 mg/kg, 8 mg/kg, 12 mg/kg, 16 mg/kg, 20 mg/kg and 27 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
  Part B: Participants received escalating doses of 8 mg/kg / 12 mg/kg / 16 mg/kg / 20 mg/kg / 27 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
  Part C: Participants received 20 mg/kg LY3127804 plus 12 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
Arm/Group | All Part A , Part B and Part C Participants
Number analyzed (Participants) | 62
milligram per kilogram (mg/kg) | 20

2. Secondary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A dose limiting toxicity (DLT) defined as an adverse event (AE) during the first 21 days that was possibly related to the study drug and fulfilled any of the following criteria using the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0: CTCAE Grade 3 nonhematologic toxicity, grade 4 neutropenia that lasted longer than 2 weeks, grade ≥3 thrombocytopenia complicated by hemorrhage, and any hematologic toxicity that caused a cycle delay of >14 days; a DLT can be declared if a participant experiences increasing toxicity during treatment.
Time Frame: Baseline through Cycle 1 (28 Day Cycle)
Population: All randomized participants who received at least one dose of study drug (ramucirumab and/or LY3127804) and had DLTs in Part A, Part B and Part C.
Measure: Number; unit: participants
Groups:
- Part B Cohort 6: 27 mg/kg LY3127804 + 8 mg/kg Ramucirumab: Participants received 27 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
Arm/Group | Part A Cohort 1: 4 mg/kg LY3127804 | Part A Cohort 2: 8 mg/kg LY3127804 | Part A Cohort 3: 12 mg/kg LY3127804 | Part A Cohort 4: 16 mg/kg LY3127804 | Part A Cohort 5: 20 mg/kg LY3127804 | Part A Cohort 6: 27 mg/kg LY3127804 | Part B Cohort 2: 8 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 3: 12 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 4: 16 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 5: 20 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 6: 27 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part C: 20 mg/kg LY3127804 +12 mg/kg Ramucirumab
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 4 | 6 | 7 | 7 | 7 | 8 | 7
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve (AUC) of LY3127804
Description: Area under the plasma concentration-time curve of LY3127804 over the dosing interval (AUC[0-τ]) from time 0 to 336 hours (h) was evaluated.
Time Frame: predose, end of infusion (1h), 2h, 24h, 96h, 168h, 336 h following dose on day 1 and at predose, end of infusion (1h), 24h, 168h and 336 h following dose on day 15 and at predose, end of infusion (1h), 2h, 168h, 336h following dose on day 29
Population: All randomized participants who received at least one dose of study drug (LY3127804) with evaluable PK data in Part A, Part B and Part C. Per protocol, similar strength doses of LY3127804 from Part A, B, and C were combined for measuring PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter(µg*hr/mL)
Groups:
- 4 mg/kg LY3127804: Participants from Part A received 4 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- 8 mg/kg LY3127804: Participants from Part A and Part B received 8 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- 12 mg/kg LY3127804: Participants from Part A and Part B received 12 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- 16 mg/kg LY3127804: Participants from Part A and Part B received 16 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- 20 mg/kg LY3127804: Participants from Part A, Part B and Part C received 20 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- 27 mg/kg LY3127804: Participants from Part A and Part B received 27 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
Arm/Group | 4 mg/kg LY3127804 | 8 mg/kg LY3127804 | 12 mg/kg LY3127804 | 16 mg/kg LY3127804 | 20 mg/kg LY3127804 | 27 mg/kg LY3127804
Number analyzed (Participants) | 3 | 9 | 9 | 10 | 17 | 12
microgram*hour per milliliter(µg*hr/mL)
  Day 1 dose: number analyzed (Participants) | 3 | 6 | 9 | 9 | 17 | 12
  Day 1 dose | 11631 (30) | 29817 (25) | 33036 (31) | 43636 (25) | 57917 (23) | 81931 (28)
  Day 15 dose: number analyzed (Participants) | 3 | 9 | 6 | 10 | 13 | 9
  Day 15 dose | 16647 (33) | 42486 (22) | 47084 (35) | 65837 (39) | 85529 (22) | 108015 (24)
  Day 29 dose: number analyzed (Participants) | 2 | 5 | 8 | 5 | 10 | 8
  Day 29 dose | 16136 (27) | 53889 (41) | 62327 (26) | 93032 (25) | 106655 (28) | 120607 (29)

4. Secondary Outcome: Pharmacokinetics: AUC of Ramucirumab in Combination With LY3127804
Description: Area under the serum concentration-time curve of ramucirumab in combination with LY3127804 over the dosing interval (AUC[0-τ]) from time 0 to 336 hours (τ) was evaluated following the first dose.
Time Frame: predose, end of infusion (1h), 24h, 96h, 168h, 336 h following Ramucirumab dose on day 1
Population: All randomized participants who received at least one dose of study drug (ramucirumab and/or LY3127804) with evaluable PK data in Part B and Part C. Per protocol, Part B reporting arms in cohorts 2 to 6 were combined to measure ramucirumab PK in presence of LY3127804.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Groups:
- Part B Cohorts 2 to 6: LY3127804 + 8 mg/kg Ramucirumab: Participants received 8 mg/kg,12 mg/kg,16 mg/kg, 20 mg/kg, 27 mg/kg LY3127804 LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
Arm/Group | Part B Cohorts 2 to 6: LY3127804 + 8 mg/kg Ramucirumab | Part C: 20 mg/kg LY3127804 +12 mg/kg Ramucirumab
Number analyzed (Participants) | 18 | 7
µg*h/mL | 20615 (32) | 35403 (16)

5. Secondary Outcome: Number of Participants With Anti-LY3127804 Antibodies
Description: The number of participants who had treatment-emergent or follow-up emergent anti-drug antibodies (ADA) is reported. Participants with treatment-emergent ADA were defined as participants who had any sample from cycle 1 pre-Dose through 30 days after last dose of study drug that was a 4-fold increase (2 dilution increase) in immunogenicity titer over the baseline titer, or participants who tested negative at baseline and positive post-baseline (at titer of ≥1:20).
Time Frame: Cycle 1 Pre-Dose through 30 Days After Last Dose of Study Drug (Up To 5 Months)
Population: All randomized participants who received at least one dose of study drug (ramucirumab and/or LY3127804) and had a baseline and at least 1 post-baseline ADA assessment in Part A, Part B and Part C.
Measure: Number; unit: participants
Arm/Group | Part A Cohort 1: 4 mg/kg LY3127804 | Part A Cohort 2: 8 mg/kg LY3127804 | Part A Cohort 3: 12 mg/kg LY3127804 | Part A Cohort 4: 16 mg/kg LY3127804 | Part A Cohort 5: 20 mg/kg LY3127804 | Part A Cohort 6: 27 mg/kg LY3127804 | Part B Cohort 2: 8 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 3: 12 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 4: 16 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 5: 20 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 6: 27 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part C: 20 mg/kg LY3127804 +12 mg/kg Ramucirumab
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 6 | 6 | 7 | 7 | 7 | 7
participants | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0

6. Secondary Outcome: Number of Participants With Anti-Ramucirumab Antibodies
Description: as for outcome 5
Time Frame: Cycle 1 Pre-Dose through 30 Days After Last Dose of Study Drug (Up to 5 Months)
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- Part A Cohort 3: 12mg/kg LY3127804: Participants received 12 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part A Cohort 4: 16mg/kg LY3127804: Participants received 16 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part A Cohort 5: LY3127804-20mg/kg: Participants received 20 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part A Cohort 6: 27mg/kg LY3127804: Participants received 27 mg/kg LY3127804 administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part B Cohort 2: 8mg/kg LY3127804 + 8mg/kg Ramucirumab: Participants received 8 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part B Cohort 3: 12mg/kg LY3127804 + 8mg/kg Ramucirumab: Participants received 12 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part B Cohort 4: 16mg/kg LY3127804 + 8mg/kg Ramucirumab: Participants received 16 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part B Cohort 5: 20mg/kg LY3127804 + 8mg/kg Ramucirumab: Participants received 20 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part B Cohort 6: 27mg/kg LY3127804 + 8mg/kg: Participants received 27 mg/kg LY3127804 plus 8 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
- Part C: 20mg/kg LY3127804 +12mg/kg Ramucirumab: Participants received 20 mg/kg LY3127804 plus 12 mg/kg ramucirumab administered as IV infusion on days 1 and 15 of a 28-day cycle.
Arm/Group | Part A Cohort 1: 4 mg/kg LY3127804 | Part A Cohort 2: 8 mg/kg LY3127804 | Part A Cohort 3: 12mg/kg LY3127804 | Part A Cohort 4: 16mg/kg LY3127804 | Part A Cohort 5: LY3127804-20mg/kg | Part A Cohort 6: 27mg/kg LY3127804 | Part B Cohort 2: 8mg/kg LY3127804 + 8mg/kg Ramucirumab | Part B Cohort 3: 12mg/kg LY3127804 + 8mg/kg Ramucirumab | Part B Cohort 4: 16mg/kg LY3127804 + 8mg/kg Ramucirumab | Part B Cohort 5: 20mg/kg LY3127804 + 8mg/kg Ramucirumab | Part B Cohort 6: 27mg/kg LY3127804 + 8mg/kg | Part C: 20mg/kg LY3127804 +12mg/kg Ramucirumab
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 6 | 6 | 7 | 7 | 7 | 7
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Who Exhibit Complete Response (CR) or Partial Response (PR) [Overall Response Rate (ORR)]
Description: ORR defined as the percentage of participants who achieve a CR or PR as assessed by RECIST v.1.1. The ORR is the number of participants with a complete response (CR) or partial response (PR) divided by the number of randomized participants recorded between the date of randomization and the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever comes first. Complete response (CR) is defined as disappearance of all target (and non-target) lesions, and normalization of tumor marker level. Partial response (PR) is defined as at least a 30% decrease in the sum of longest diameters of target lesions, taking as reference the baseline sum of longest diameters.
Time Frame: Baseline through Measured Progressive Disease or Death (Up to 4 Months)
Population: All randomized participants who had adequate baseline and at least 1 post-baseline tumor assessments in Part A, Part B and Part C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A Cohort 1: 4 mg/kg LY3127804 | Part A Cohort 2: 8 mg/kg LY3127804 | Part A Cohort 3: 12 mg/kg LY3127804 | Part A Cohort 4: 16 mg/kg LY3127804 | Part A Cohort 5: 20 mg/kg LY3127804 | Part A Cohort 6: 27 mg/kg LY3127804 | Part B Cohort 2: 8 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 3: 12 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 4: 16 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 5: 20 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 6: 27 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part C: 20 mg/kg LY3127804 +12 mg/kg Ramucirumab
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 4 | 6 | 7 | 7 | 7 | 8 | 7
percentage of participants | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 60.2] | 33.3 [4.3 to 77.7] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 41.0] | 12.5 [0.3 to 52.7] | 14.3 [0.4 to 57.9]

8. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) time is defined as the time from the date of randomization to the first date of documented objective progressive disease (PD) or death from any cause. For participants who were not known to have had objective PD as of the data inclusion cut-off date for a particular analysis, PFS was censored at the date of the last objective progression-free disease assessments. For participants who took any subsequent systemic anticancer therapy prior to progression, PFS was censored at the date of the last objective progression-free disease assessment prior to the start date of any subsequent systemic anticancer therapy.
Time Frame: Baseline to Measured Progressive Disease or Death (Up to 4 Months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A Cohort 1: 4 mg/kg LY3127804 | Part A Cohort 2: 8 mg/kg LY3127804 | Part A Cohort 3: 12 mg/kg LY3127804 | Part A Cohort 4: 16 mg/kg LY3127804 | Part A Cohort 5: 20 mg/kg LY3127804 | Part A Cohort 6: 27 mg/kg LY3127804 | Part B Cohort 2: 8 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 3: 12 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 4: 16 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 5: 20 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 6: 27 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part C: 20 mg/kg LY3127804 +12 mg/kg Ramucirumab
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 4 | 6 | 7 | 7 | 7 | 8 | 7
Months | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Baseline Up to 54 Months
Description: All randomized participants in Part A, Part B and Part C.
Arm/Group | Part A Cohort 1: 4 mg/kg LY3127804 | Part A Cohort 2: 8 mg/kg LY3127804 | Part A Cohort 3: 12 mg/kg LY3127804 | Part A Cohort 4: 16 mg/kg LY3127804 | Part A Cohort 5: 20 mg/kg LY3127804 | Part A Cohort 6: 27 mg/kg LY3127804 | Part B Cohort 2: 8 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 3: 12 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 4: 16 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 5: 20 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part B Cohort 6: 27 mg/kg LY3127804 + 8 mg/kg Ramucirumab | Part C: 20 mg/kg LY3127804 +12 mg/kg Ramucirumab
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 1/3 | 0/3 | 1/3 | 2/4 | 0/6 | 1/7 | 2/7 | 2/7 | 3/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/3 | 1/3 | 0/3 | 2/4 | 2/6 | 2/7 | 3/7 | 3/7 | 2/8 | 5/7
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 3/3 | 3/3 | 4/4 | 6/6 | 5/7 | 7/7 | 7/7 | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: 4 mg/kg LY3127804 (N=3) | Part A Cohort 2: 8 mg/kg LY3127804 (N=4) | Part A Cohort 3: 12 mg/kg LY3127804 (N=3) | Part A Cohort 4: 16 mg/kg LY3127804 (N=3) | Part A Cohort 5: 20 mg/kg LY3127804 (N=3) | Part A Cohort 6: 27 mg/kg LY3127804 (N=4) | Part B Cohort 2: 8 mg/kg LY3127804 + 8 mg/kg Ramucirumab (N=6) | Part B Cohort 3: 12 mg/kg LY3127804 + 8 mg/kg Ramucirumab (N=7) | Part B Cohort 4: 16 mg/kg LY3127804 + 8 mg/kg Ramucirumab (N=7) | Part B Cohort 5: 20 mg/kg LY3127804 + 8 mg/kg Ramucirumab (N=7) | Part B Cohort 6: 27 mg/kg LY3127804 + 8 mg/kg Ramucirumab (N=8) | Part C: 20 mg/kg LY3127804 +12 mg/kg Ramucirumab (N=7)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: 4 mg/kg LY3127804 (N=3) | Part A Cohort 2: 8 mg/kg LY3127804 (N=4) | Part A Cohort 3: 12 mg/kg LY3127804 (N=3) | Part A Cohort 4: 16 mg/kg LY3127804 (N=3) | Part A Cohort 5: 20 mg/kg LY3127804 (N=3) | Part A Cohort 6: 27 mg/kg LY3127804 (N=4) | Part B Cohort 2: 8 mg/kg LY3127804 + 8 mg/kg Ramucirumab (N=6) | Part B Cohort 3: 12 mg/kg LY3127804 + 8 mg/kg Ramucirumab (N=7) | Part B Cohort 4: 16 mg/kg LY3127804 + 8 mg/kg Ramucirumab (N=7) | Part B Cohort 5: 20 mg/kg LY3127804 + 8 mg/kg Ramucirumab (N=7) | Part B Cohort 6: 27 mg/kg LY3127804 + 8 mg/kg Ramucirumab (N=8) | Part C: 20 mg/kg LY3127804 +12 mg/kg Ramucirumab (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hypocoagulable state (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 2 (2) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (3) | 1 (1) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (4) | 4 (4) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (6) | 2 (3) | 3 (5) | 4 (6) | 4 (4) | 2 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deficiency of bile secretion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 3 (4) | 1 (1) | 1 (6) | 2 (2)
Hemianopia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (6) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (4) | 2 (4) | 2 (2) | 4 (13) | 3 (6) | 4 (9)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
No participants were enrolled in Part D and Part E reporting arms as these were deleted from protocol last amendment (based on the primary and secondary outcomes/ results of Part A-C).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT02597036/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT02597036/SAP_001.pdf